CLINICAL TRIAL: NCT01992185
Title: Pilot Study of Novel Topical Drug (Photocil) for the Treatment of Vitiligo
Brief Title: Photocil (Topical) for the Treatment of Vitiligo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Biology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB-DRUG-PHOTOCIL-VT-001
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Results first posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-02

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Photocil for Vitiligo (Active Comparator): Active Drug - Photocil for Vitiligo
  Interventions: Drug: Photocil for Vitiligo
- Placebo - Sunscreen (SPF 2) (Placebo Comparator): Placebo - Sunscreen (SPF 2)
  Interventions: Other: Placebo - Sunscreen (SPF 2)

INTERVENTIONS:
Drug: Photocil for Vitiligo — Photocil for Vitiligo
  Other Names: Photocil for Vitiligo (U.S. FDA NDC: 54841-001-01)
  Arms: Photocil for Vitiligo
Other: Placebo - Sunscreen (SPF 2) — Placebo - Sunscreen (SPF 2)
  Arms: Placebo - Sunscreen (SPF 2)

SUMMARY:
Photocil is a topical drug (cream) that selectively delivers Narrow Band - Ultraviolet B (NB-UVB) therapy when exposed to sunlight. Photocil is intended to help protect users from non-therapeutic Ultraviolet B (UVB) radiation while selectively passing wavelengths of light in the NB-UVB range with peak transmission of 308nm. The aim of the study is to assess the safety and efficacy of Photocil in the treatment of vitiligo.

DETAILED DESCRIPTION:
NB-UVB phototherapy is a common treatment for patients with psoriasis, and has been reported to be safe and effective in numerous clinical trials. Clinical trials have reported achievement of Vitiligo Area Severity Index (VASI)-75 in 50-70% of patients after 4-6 weeks of NB-UVB treatment.

Many drawbacks limit patients compliance, access, and acceptance of traditional NB-UVB phototherapy. The strict treatment regimen (2-3 sessions per week for an average of 12 weeks or more) performed at a specialized phototherapy clinic combined with high cost and low or no reimbursement make compliance and access a major drawback.

In order to address the drawbacks of phototherapy, we developed a novel topical cream - Photocil - that selectively delivers NB-UVB therapy when exposed to sunlight. When used with natural sunlight, Photocil provides a convenient alternative to traditional clinic based phototherapy; thus, has the potential to dramatically increase patient compliance and treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with vitiligo confirmed by a dermatologist
* Vitiligo lesions affecting at a minimum 5% of the facial, legs, or arms surface area
* Age: 18 to 65
* Participants able to give informed consent

Exclusion Criteria:

* Subject did not respond to prior phototherapy treatment
* Subject completed phototherapy for same lesion(s) in last 6 months
* Subject has previous history of skin cancer
* Subject has previous history of photosensitivity
* Subject has a history of herpes (HSV I or II) outbreaks
* Subject has previous history of autoimmune disease may be excluded at investigator's discretion
* Subject is currently taking of immunosuppressive or photosensitizing drugs
* Subject plans to use antibiotics, anti-fungal, calcineurin inhibitors or other drugs that may cause photosensitivity during the study period. These patients may be excluded at investigator's discretion
* Subject is pregnant or lactating women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McCoy, PhD, Study Director — Applied Biology, Inc.
Locations (1):
- Physicians Institute, Tucson, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Photocil for Vitiligo | Placebo - Sunscreen (SPF 2)
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Photocil for Vitiligo | Placebo - Sunscreen (SPF 2) | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (13.4) | 35.1 (15.2) | 36.5 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percent Repigmentation
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: Percent Repigmentation
Arm/Group | Photocil for Vitiligo | Placebo - Sunscreen (SPF 2)
Number analyzed (Participants) | 7 | 8
Percent Repigmentation | 48.5 (16.8) | 2.5 (7.1)

ADVERSE EVENTS:
Arm/Group | Photocil for Vitiligo | Placebo - Sunscreen (SPF 2)
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days